CLINICAL TRIAL: NCT04247230
Title: An Open Label, Placebo and Positive Controlled, Randomised, Cross-over Study in Healthy Male Volunteers to Determine the Effect on Penile Skin Sensation of a Newly Formulated Tetracaine Product PET500
Brief Title: Study to Determine the Effect of a Newly Formulated Tetracaine Product PET500 on Penile Skin Sensation
Acronym: FM48
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: FM48
Record Dates: First submitted 2019-12-14; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tetracaine; Menogaril

STUDY DESIGN:
Intervention Model Description: Von Frey hair (monofilaments) was used to assess the changes in touch sensitivity on the glans penis after the application of IMP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PET500 (0.1%) (Experimental): Each actuation of the pump spray dispenses 130µl PET500. Two pumps will dispense 260µl as follows:
  PET500 (0.1%) corresponding to a tetracaine total dose of 0.26mg
  Interventions: Drug: Tetracaine
- PET500 (0.25%) (Experimental): Each actuation of the pump spray dispenses 130µl PET500. Two pumps will dispense 260µl as follows:
  PET500 (0.25%) corresponding to a tetracaine total dose of 0.65mg
  Interventions: Drug: Tetracaine
- PET500 (0.5%) (Experimental): Each actuation of the pump spray dispenses 130µl PET500. Two pumps will dispense 260µl as follows:
  PET500 (0.5%) corresponding to a tetracaine total dose of 1.3mg
  Interventions: Drug: Tetracaine
- PET500 placebo comparator (Experimental): Each actuation of the pump spray dispenses 130µl PET500 [vehicle only]. Two pumps will dispense 260µl
  Interventions: Other: Matching placebo (PET500)
- STUD100 (9.6%) (Active Comparator): Each actuation of the pump spray dispenses 130µl, corresponding to a dose of 7.7mg lidocaine. Three pumps will dispense 390µl of a 9.6% solution, delivering a total dose of 23mg lidocaine. UK License Number PL/2294/5000R
  Interventions: Drug: STUD100

INTERVENTIONS:
Drug: Tetracaine — Von Frey hair (monofilaments) was used to assess the changes in touch sensitivity on the glans penis after the application of IMP.
  Other Names: PET500 tetracaine spray
  Arms: PET500 (0.1%); PET500 (0.25%); PET500 (0.5%)
Other: Matching placebo (PET500) — Von Frey hair (monofilaments) was used to assess the changes in touch sensitivity on the glans penis after the application of IMP.
  Other Names: PET500 Matching Placebo
  Arms: PET500 placebo comparator
Drug: STUD100 — Von Frey hair (monofilaments) was used to assess the changes in touch sensitivity on the glans penis after the application of IMP.
  Other Names: STUD100 desensitizing spray for men
  Arms: STUD100 (9.6%)

SUMMARY:
An open label, placebo and positive controlled, randomised, cross-over study in healthy male volunteers to determine the effect on penile skin sensation of a newly formulated tetracaine product PET500

DETAILED DESCRIPTION:
This was an open label, placebo and positive controlled, randomised, dose-ranging, cross-over pilot study.

On each dosing day the subjects each received one dose of tetracaine (0.26 or 0.65 or 1.3mg), or placebo, or Stud100® (which served as a positive control) on the glans penis The doses of PET500 were applied in liquid spray form (260μl) at approximately the same time of the day as the previous application to locations on the glans penis in a randomised fashion.

Von Frey hair (monofilaments) was used to assess the changes in touch sensitivity on the glans penis after the application of IMP.

The first two volunteers included in the trial piloted the sensitivity assessments prior to the inclusion of all other subjects. Changes could be made to the assessment times on the basis of the pilot data to ensure subsequent timings were relevant. However any such changes were not to expose volunteers to more assessments than were specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male healthy subject aged 18 to 65 years, inclusive.
2. The subject is capable of understanding and complying with protocol requirements.
3. The subject is in good health as determined by medical history and physical examination at screening.
4. The subject signs a written, informed consent form prior to the initiation of any study procedures

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1 History or hypersensitivity to tetracaine or ethanol.

2. History or signs of a sexually transmitted disease.

3. Any current penile abnormalities.

4. Known current drug abuser or alcoholic as determined by medical history.

5. Participation in a clinical trial within the last month prior to dosing on Day 1.

6. The use of concomitant systemic or topical medications or foods that may affect the study outcome and / or impair drug metabolising capacity.

7. A positive HIV 1 & 2 antibodies, Hepatitis B surface antigen, and/or Hepatitis C antibody result.

8. Unfit to participate in the study in the opinion of the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2008-10-20 (Actual); Study Completion 2009-02-23 (Actual)

PRIMARY OUTCOMES:
Onset of action of different doses of a newly formulated tetracaine spray PET500 when applied to the glans penis assessed using Von Frey fibres (monofilaments) to measure touch sensitivity | 2 Months
  To determine the onset of action of different doses of a newly formulated tetracaine spray PET500 when applied to the glans penis (compared to placebo and positive prilocaine/lidocaine control).
Duration of action of different doses of a newly formulated tetracaine spray PET500 when applied to the glans penis using Von Frey fibres (monofilaments) to measure touch sensitivity | 2 Months
  To determine the duration of action of different doses of a newly formulated tetracaine spray PET500 when applied to the glans penis (compared to placebo and positive prilocaine/lidocaine control).

SECONDARY OUTCOMES:
Incidence of adverse events for PET500 | 2 months
  To determine incidence, of adverse events by Treatment group for doses of a newly formulated tetracaine spray PET500 in healthy male volunteers.
Intensity and relationship of adverse events to PET500 | 2 months
  To determine intensity and relationship to study drug of adverse events by Treatment group for doses of a newly formulated tetracaine spray PET500 in healthy male volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, Dr, Principal Investigator — Richmond Pharmacology

IPD SHARING:
Plan to Share IPD: No